CLINICAL TRIAL: NCT01620216
Title: A Phase II Proof-of-Concept Trial to Study Kinase Inhibition in Relapsed/Refractory Acute Leukemias: Using a Comprehensive In Vitro Kinase Inhibitor Panel to Select Individualized, Targeted Therapies
Brief Title: Targeted Therapy in Treating Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia or Acute Myelogenous Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit enough eligible subjects
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Stephen Spurgeon, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00007195; NCI-2012-01084 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CA180-392; IRB00007195 (Other: OHSU Knight Cancer Institute); R21CA159265 (NIH)
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Results first posted 2021-10-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia; Recurrent Acute Lymphoblastic Leukemia; Recurrent Acute Myeloid Leukemia; Refractory Acute Lymphoblastic Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Drug Screening Assays, Antitumor; Dasatinib; idelalisib; 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; ponatinib; ruxolitinib; Sorafenib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Group I (dasatinib) (Experimental): Patients receive dasatinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Antitumor Drug Screening Assay; Drug: Dasatinib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Group II (sutinib malate) (Experimental): Patients receive sutinib malate PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Antitumor Drug Screening Assay; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sunitinib; Drug: Sunitinib Malate
- Group III (sorafenib tosylate) (Experimental): Patients receive sorafenib tosylate PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Antitumor Drug Screening Assay; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sorafenib; Drug: Sorafenib Tosylate
- Group IV (ponatinib hydrochloride) (Experimental): Patients receive ponatinib hydrochloride PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity
  Interventions: Other: Antitumor Drug Screening Assay; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Ponatinib; Drug: Ponatinib Hydrochloride
- Group V (pacritinib) (Experimental): Patients receive pacritinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Antitumor Drug Screening Assay; Other: Laboratory Biomarker Analysis; Drug: Pacritinib; Other: Pharmacological Study
- Group VI (ruxolitinib) (Experimental): Patients receive ruxolitinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Antitumor Drug Screening Assay; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Ruxolitinib
- Group VII (idelalisib) (Experimental): Patients receive idelalisib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Antitumor Drug Screening Assay; Drug: Idelalisib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Other: Antitumor Drug Screening Assay — Undergo pre clinical kinase inhibitor activity screening
  Other Names: Drug Screening Assays, Antitumor
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
  Arms: Group I (dasatinib)
Drug: Idelalisib — Given PO
  Other Names: CAL-101; GS 1101; GS-1101; Phosphoinositide-3 Kinase Delta Inhibitor CAL-101; Zydelig
  Arms: Group VII (idelalisib)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pacritinib — Given PO
  Other Names: Oral JAK2 Inhibitor SB1518; SB 1518; SB-1518; SB1518
  Arms: Group V (pacritinib)
Other: Pharmacological Study — Correlative studies
Drug: Ponatinib — Given PO
  Other Names: AP-24534; AP24534
  Arms: Group IV (ponatinib hydrochloride)
Drug: Ponatinib Hydrochloride — Given PO
  Other Names: AP24534 HCl; Iclusig
  Arms: Group IV (ponatinib hydrochloride)
Drug: Ruxolitinib — Given PO
  Other Names: INCB-18424; INCB18424; Jakafi; Oral JAK Inhibitor INCB18424
  Arms: Group VI (ruxolitinib)
Drug: Sorafenib — Given PO
  Other Names: BA4 43 9006; BAY 43-9006; Bay-439006
  Arms: Group III (sorafenib tosylate)
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib
  Arms: Group III (sorafenib tosylate)
Drug: Sunitinib — Given PO
  Arms: Group II (sutinib malate)
Drug: Sunitinib Malate — Given PO
  Other Names: SU011248; SU11248; sunitinib; Sutent
  Arms: Group II (sutinib malate)

SUMMARY:
This phase II trial studies how well targeted therapy works in treating patients with acute lymphoblastic leukemia or acute myelogenous leukemia that has come back after a period of improvement or does not respond to treatment. Testing patients' blood or bone marrow to find out if their type of cancer may be sensitive to a specific drug may help doctors choose more effective treatments. Dasatinib, sunitinib malate, sorafenib tosylate, ponatinib hydrochloride, pacritinib, ruxolitinib, and idelalisib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving targeted therapy based on cancer type may be an effective treatment for acute lymphoblastic leukemia or acute myelogenous leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the clinical activity of kinase inhibitors using pre-clinical (in-vitro) activity to select individual therapy.

SECONDARY OBJECTIVES:

I. To evaluate overall objective response rates (complete response plus partial response).

II. Determine overall survival (OS) and progression-free survival (PFS).

EXPLORATORY/CORRELATIVE OBJECTIVES:

I. Prioritize active/aberrant kinase pathways using an in vitro inhibitor screen using individual primary leukemia samples.

II. Measure "on target" in vivo kinase inhibition and signal transducer and activator of transcription (STAT)-5 phosphorylation and correlate with response to treatment.

III. Perform next generation sequencing (whole exome sequencing) for complete mutational analysis.

IV. Identify aberrant gene expression in primary leukemia samples from study subjects.

V. Evaluate pharmacokinetics for each individual kinase inhibitor during therapy.

OUTLINE: Patients are assigned to 1 of 7 treatment groups based on pre-clinical kinase inhibitor activity.

GROUP I: Patients receive dasatinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive sutinib malate PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

GROUP III: Patients receive sorafenib tosylate PO twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

GROUP IV: Patients receive ponatinib hydrochloride PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

GROUP V: Patients receive pacritinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

GROUP VI: Patients receive ruxolitinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

GROUP VII: Patients receive idelalisib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Participants >= 18 years of age with relapsed/refractory leukemia with a confirmed diagnosis of acute myelogenous leukemia (AML) or acute lymphoblastic leukemia (ALL) who meet the following criteria:

  * Individuals aged 18-64 years with salvage treatment failures only - defined as relapsed or refractory to after least 1 cycle of salvage therapy

    * Given the clinical activity and use of hypomethylating agents in AML patients, initial and salvage therapy may include hypomethylating agents
  * Age >= 65 years: Refractory to induction chemotherapy - defined as no response to initial therapy or have relapsed after initial therapy

    * Individuals aged >= 65 years, with chronic myelomonocytic leukemia (CMML) or myelodysplasia (MDS) that transform to acute leukemia while actively receiving hypomethylating agents (i.e., decitabine or azacytidine) will be considered induction failures and are thus eligible for this trial; for Philadelphia positive (Ph+) ALL, initial therapy and salvage therapy may include steroids and imatinib or dasatinib
* Primary patient samples must show in vitro kinase inhibitor sensitivity as determined by the Oregon Health and Science University (OHSU) functional kinase inhibitor screen; for OHSU patients, functional kinase inhibitor screening may be performed as part of this study or through enrollment in eIRB4422 if the identical Food and Drug Administration (FDA)/Clinical Laboratory Improvement Act (CLIA) approved assay is used and a result is available within 2 weeks of starting on study drug treatment
* Patients must have normal organ function as defined below:

  * Serum creatinine < 2.0 x institutional upper limit of normal (ULN)
  * International normalized ratio (INR) < 1.5 x institutional ULN
* Adequate hepatic function as defined by the following criteria:

  * Total serum bilirubin =< 1.5 x ULN, unless due to Gilbert's syndrome
  * Alanine aminotransferase (ALT) =< 2.5 x ULN
  * Aspartate aminotransferase (AST) =< 2.5 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Discontinuation of anti-coagulants and anti-platelet drugs at least 7 days prior to start of study drug

  * Aspirin 81 mg is permitted as long as platelet count is > 50 and there is no evidence of active bleeding or coagulopathy (INR > 1.5, fibrinogen > 150)
* No uncontrolled infections as determined by the investigator
* No clinically significant thyroid disease (e.g. hyperthyroid/hypothyroidism)
* No active graft versus host disease (GVHD): patients with a history of stem cell transplant are eligible but cannot have evidence of active GVHD as determined by the investigator
* Must be able to take oral medication
* Women of childbearing potential must have a negative serum or urine pregnancy test (sensitivity < 25 IU human chorionic gonadotropin [HCG]/L) within 72 hours prior to the start of study drug
* Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped; women of childbearing potential and men with a sexual partner of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy
* Ability to understand and the willingness to sign a written informed consent and Health Insurance Portability and Accountability Act (HIPPA) document
* Serum sodium (Na), potassium (K), magnesium (Mg), and total serum calcium (Ca) or ionized Ca levels must be greater than or equal to the institutional lower limit of normal; subjects with low K or Mg levels, total corrected serum Ca and/or ionized Ca must be replete for protocol entry
* Dasatinib

  * Discontinuation of any medications known to contribute significantly to the risk of QT prolongation at least 48 hours prior to start of study drug; Levaquin and Zofran are an exception; of note, certain agents that prolong the corrected QT (QTc) may be allowed but only after discussion with the chemotherapy pharmacist; should the investigator believe that therapy with a potentially QT prolonging medication is vital to an individual subject's care, then additional electrocardiogram (ECG)s should be done at the investigator's discretion to ensure the subject's safety
  * Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug
  * Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 90 days (duration of sperm turnover) for a total of 90 days post-treatment completion
  * Azoospermic males and WOCBP, who are not heterosexually active, are exempt from contraceptive requirements; however, WOCBP must still under pregnancy testing as described in this section
  * Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of unexpected pregnancy; investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective contraception; highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly
  * At a minimum, subjects must agree to the use of two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective
* Sorafenib

  * Creatinine < 1.5 X ULN
* Ponatinib

  * Female and male patients who are fertile must agree to use an effective form of contraception with their sexual partners from randomization through 4 months after the end of treatment
  * Discontinuation of any medications known to contribute significantly to the risk of QT prolongation at least 48 hours prior to start of study drug; Levaquin and Zofran are an exception; of note, certain agents that prolong the QTc may be allowed but only after discussion with the chemotherapy pharmacist; should the investigator believe that therapy with a potentially QT prolonging medication is vital to an individual subject's care, then additional ECGs should be done at the investigator's discretion to ensure the subject's safety
  * Serum lipase =< 1.5 x ULN
  * Serum amylase =< 1.5 x ULN
* Pacritinib

  * Discontinuation of any medications known to contribute significantly to the risk of QT prolongation at least 48 hours prior to start of study drug; Levaquin and Zofran are an exception; of note, certain agents that prolong the QTc may be allowed but only after discussion with the chemotherapy pharmacist; should the investigator believe that therapy with a potentially QT prolonging medication is vital to an individual subject's care, then additional ECGs should be done at the investigator's discretion to ensure the subject's safety

Exclusion Criteria:

* Any leukemia treatment within 1 week (for cytotoxic therapy) and/or 5 half lives (for targeted agents) prior to starting study drug; corticosteroids are allowable throughout the study to treat concomitant medical disorders per provider discretion; hydroxyurea is allowed prior to enrollment and after the start of the study drug for the control of peripheral leukemic blasts in subjects with leukocytosis per physician discretion
* Recent uncontrolled angina, recent > New York Heart Association (NYHA) class II congestive heart failure, or recent myocardial infarction (MI) within 6 months prior to start of study treatment
* Diagnosed congenital long QT syndrome
* Any recent history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
* History of clinically significant bleeding disorder unrelated to cancer
* Drugs that affect the cytochrome P450 family 3 subfamily A polypeptide 4 (CYP3A4) system (inducers/inhibitors/substrates) are allowed but should be used with caution depending on specific kinase inhibitor used; dietary supplements will be discouraged; however, their use may be allowed on a case by case basis per the discretion of the investigator after consultation with an oncology pharmacist
* Uncontrolled intercurrent illness that would limit compliance with study requirements
* Pregnant or lactating women are excluded from this study
* Known human immunodeficiency virus (HIV)-positive patients are excluded from the study
* History of hypersensitivity to any of the kinase inhibitors included in this study
* Dasatinib

  * Known pulmonary arterial hypertension
  * Patients may not have a clinically significant pleural or pericardial effusion
  * Uncontrolled hypertension: inability to maintain blood pressure below the limit of 140/90 mmHg
  * Any history of second or third degree heart block (may be eligible if the subject currently has a pacemaker)
  * Prolonged QTc interval (> 450 msec for men and > 470 msec for women) on pre-entry electrocardiogram
* Sorafenib

  * Major surgery, open biopsy, or significant traumatic injury within 30 days
  * Non-healing wound, ulcer, or bone fracture
  * Thrombotic or embolic venous or arterial events, such as cerebrovascular accident, including transient ischemic attacks, arterial thrombosis, deep vein thrombosis and pulmonary embolism within the past 6 months

    * Line associated deep vein thrombosis (DVTs) which are adequately treated (line removed and/or patient anticoagulated) are permitted
  * Uncontrolled hypertension
  * Active bleeding during screening
* Ponatinib

  * History of acute pancreatitis within 1 year of study or history of chronic pancreatitis
  * QTC > 450 msec for men and > 470 msec for women
  * Uncontrolled hypertriglyceridemia (triglycerides > 450 mg/dL)
  * Any history of myocardial infarction, stroke, or revascularization
  * Any history of venous thromboembolism including deep venous thrombosis or pulmonary embolism
  * Unstable angina or transient ischemic attack within 6 months prior to start of study treatment
  * Congestive heart failure within 6 months prior to enrollment, or left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards within 6 months prior to enrollment
  * History of clinically significant (as determined by the treating physician) atrial arrhythmia
  * Uncontrolled hypertension (diastolic blood pressure > 90 mm Hg; systolic > 140 mm Hg); patients with hypertension should be under treatment on study entry to effect blood pressure control
  * History of ongoing alcohol abuse
  * Ocular toxicity present as measure during a comprehensive eye exam
* Pacritinib

  * Major surgery, open biopsy, or significant traumatic injury within 30 days
  * Active bleeding during screening
  * QTC > 450 mSec for men and > 470 msec for women
  * NYHA class II congestive heart failure (a history of CHF is allowed as long as this has resolved to < NYHA class II within 30 days of initiation of pacritinib
* Ruxolitinib

  * Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or risk of reactivation: HBV deoxyribonucleic acid (DNA) and HCV ribonucleic acid (RNA) must be undetectable; subjects cannot be positive for hepatitis B surface antigen (HBsAg) or anti-hepatitis B core antibody; subjects who have positive anti-hepatitis B surface antibdy (HBs) as the only evidence of prior exposure may participate in the study provided that there is both 1) no known history of HBV infection, and 2) verified receipt of hepatitis B vaccine
* Idelalisib

  * Ongoing drug-induced liver injury, chronic active hepatitis C (HCV), chronic active hepatitis B (HBV), alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, portal hypertension, or history of autoimmune hepatitis
  * Ongoing symptomatic pneumonitis.
  * Ongoing inflammatory bowel disease or autoimmune colitis.
  * Ongoing cytomegalovirus (CMV) infection, treatment, or prophylaxis within the past 28 days prior to the screening test for active CMV
  * History of serious allergic reaction including anaphylaxis and epidermal necrolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05-11 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Loriaux, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I (Dasatinib) | Group II (Sutinib Malate) | Group III (Sorafenib Tosylate) | Group IV (Ponatinib Hydrochloride) | Group V (Pacritinib) | Group VI (Ruxolitinib) | Group VII (Idelalisib)
Started | 4 | 2 | 6 | 0 | 0 | 0 | 0
Completed | 4 | 2 | 6 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Zero patients were enrolled in the Ponatinib, Pacritinib, Ruxolitinib, and Idealisib arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Dasatinib) | Group II (Sutinib Malate) | Group III (Sorafenib Tosylate) | Group IV (Ponatinib Hydrochloride) | Group V (Pacritinib) | Group VI (Ruxolitinib) | Group VII (Idelalisib) | Total
Number analyzed (Participants) | 4 | 2 | 6 | 0 | 0 | 0 | 0 | 12
Age, Continuous [Median (Full Range); unit: Years] | 70.5 [69 to 74] | 50 [47 to 53] | 57.5 [31 to 72] |  |  |  |  | 63 [31 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 5 |  |  |  |  | 7
  Male | 3 | 1 | 1 |  |  |  |  | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 3 | 2 | 4 |  |  |  |  | 9
  Race/Ethnicity: Hispanic or Latino | 1 | 0 | 2 |  |  |  |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Clinical Activity
Description: Will be defined as defined as a decrease of at least 25% in bone marrow blast counts or peripheral blood blast. The proportion of patients achieving the endpoint along with its 95% exact binomial confidence interval will be presented.
Time Frame: Up to 28 days
Population: Zero patients enrolled in Ponatinib, Pacrtitinib, Ruxolitinib, and Idealisib arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Dasatinib) | Group II (Sutinib Malate) | Group III (Sorafenib Tosylate) | Group IV (Ponatinib Hydrochloride) | Group V (Pacritinib) | Group VI (Ruxolitinib) | Group VII (Idelalisib)
Number analyzed (Participants) | 4 | 2 | 6 | 0 | 0 | 0 | 0
Participants | 1 | 0 | 4 |  |  |  |

2. Secondary Outcome: Overall Objective Response Rates (Complete and Partial)
Description: Per Response Evaluation Criteria in AML or ALL: Complete Response (CR), at least <5% bone marrow blasts; Partial Response (PR), reduction of >=50% bone marrow blasts; Overall Response (OR)= CR + PR.
  The proportion of patients achieving the endpoint along with its 95% exact binomial confidence interval will be presented.
Time Frame: Up to 3 years
Population: Zero patients enrolled in Ponatinib, Pacritinib, Ruxolitinib, and Idealisib arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Dasatinib) | Group II (Sutinib Malate) | Group III (Sorafenib Tosylate) | Group IV (Ponatinib Hydrochloride) | Group V (Pacritinib) | Group VI (Ruxolitinib) | Group VII (Idelalisib)
Number analyzed (Participants) | 4 | 2 | 6 | 0 | 0 | 0 | 0
Participants
  Partial response | 0 | 0 | 1 |  |  |  |
  Progressive disease | 2 | 0 | 0 |  |  |  |
  Stable disease | 2 | 2 | 4 |  |  |  |
  Not assessable | 0 | 0 | 1 |  |  |  |

3. Secondary Outcome: Progression-free Survival
Description: Kaplan-Meier method will be used to estimate the survival curve.
Time Frame: From the start of study drug treatment to death, regardless of cause of death, or date of disease progression defined as a >= 50% increase in leukemic bone marrow blasts, whichever occurs first, assessed up to 3 years
Population: Zero patients enrolled in Ponatinib, Pacritinib, Ruxolitinib, and Idealisib arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Dasatinib) | Group II (Sutinib Malate) | Group III (Sorafenib Tosylate) | Group IV (Ponatinib Hydrochloride) | Group V (Pacritinib) | Group VI (Ruxolitinib) | Group VII (Idelalisib)
Number analyzed (Participants) | 4 | 2 | 6 | 0 | 0 | 0 | 0
Participants | 1 | 1 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Overall Survival
Description: Kaplan-Meier method will be used to estimate the survival curve.
Time Frame: From the date of subject registration to death, regardless of causes of death, assessed up to 3 years
Population: Zero patients enrolled in Ponatinib, Pacritinib, Ruxolitinib, and Idealisib arms.
Measure: Mean (Full Range); unit: Days
Arm/Group | Group I (Dasatinib) | Group II (Sutinib Malate) | Group III (Sorafenib Tosylate) | Group IV (Ponatinib Hydrochloride) | Group V (Pacritinib) | Group VI (Ruxolitinib) | Group VII (Idelalisib)
Number analyzed (Participants) | 4 | 2 | 6 | 0 | 0 | 0 | 0
Days | 57 [18 to 147] | 75 [6 to 144] | 130 [43 to 430] |  |  |  |

5. Secondary Outcome: Clinical Activity
Description: Will be defined as a decrease of at least 25% in bone marrow blast counts or in peripheral blood blasts in subjects who have failed the initial inhibitor but are then treated with another inhibitor identified on repeat pre-clinical activity testing. The proportion of patients achieving the endpoint along with its 95% exact binomial confidence interval will be presented.
Time Frame: Up to 28 days
Population: Zero patients enrolled in Ponatinib, Pacritinib, Ruxolitinib, and Idealisib arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Dasatinib) | Group II (Sutinib Malate) | Group III (Sorafenib Tosylate) | Group IV (Ponatinib Hydrochloride) | Group V (Pacritinib) | Group VI (Ruxolitinib) | Group VII (Idelalisib)
Number analyzed (Participants) | 4 | 2 | 6 | 0 | 0 | 0 | 0
Participants | 0 | 0 | 0 |  |  |  |

6. Other Pre Specified Outcome: Presence of Active/Aberrant Kinase Pathways
Description: Presence of active/aberrant kinase pathways will be determined using a small molecule kinase inhibitor screen, to rapidly identify therapeutic tyrosine kinase targets in leukemia patients while simultaneously providing individualized therapeutic options. Will be correlated with treatment response, mutational analysis using next generation sequencing, and characterization of aberrant gene expression in primary leukemia samples.
Time Frame: Up to 3 years
Population: Zero patients enrolled in Ponatinib, Pacritinib, Ruxolitinib, and Idealisib arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Dasatinib) | Group II (Sutinib Malate) | Group III (Sorafenib Tosylate) | Group IV (Ponatinib Hydrochloride) | Group V (Pacritinib) | Group VI (Ruxolitinib) | Group VII (Idelalisib)
Number analyzed (Participants) | 4 | 2 | 6 | 0 | 0 | 0 | 0
Participants | 4 | 2 | 6 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection began on the first day of the start of the induction chemotherapy and continued until 30 days post last dose of study drug.
Description: Zero patients enrolled in Ponatinib, Pacritinib, Ruxolitinib, and Idealisib arms.
Groups:
- Group II (Sunitinib Malate): Patients receive sutinib malate PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Antitumor Drug Screening Assay: Undergo pre clinical kinase inhibitor activity screening
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Sunitinib: Given PO
  Sunitinib Malate: Given PO
Arm/Group | Group I (Dasatinib) | Group II (Sunitinib Malate) | Group III (Sorafenib Tosylate) | Group IV (Ponatinib Hydrochloride) | Group V (Pacritinib) | Group VI (Ruxolitinib) | Group VII (Idelalisib)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2 | 0/6 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/2 | 5/6 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/4 | 0/2 | 6/6 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Dasatinib) (N=4) | Group II (Sunitinib Malate) (N=2) | Group III (Sorafenib Tosylate) (N=6) | Group IV (Ponatinib Hydrochloride) (N=0) | Group V (Pacritinib) (N=0) | Group VI (Ruxolitinib) (N=0) | Group VII (Idelalisib) (N=0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | NA | NA | NA | NA
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | NA | NA | NA | NA
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA | NA
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA | NA
Febrile neutropenia (Investigations) | 0 (0) | 0 (0) | 4 (5) | NA | NA | NA | NA
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA | NA
Hypoalbumenia (Metabolism and nutrition disorders) | 0 | 0 (0) | 1 (1) | NA | NA | NA | NA
Lipase increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA | NA
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Dasatinib) (N=4) | Group II (Sunitinib Malate) (N=2) | Group III (Sorafenib Tosylate) (N=6) | Group IV (Ponatinib Hydrochloride) (N=0) | Group V (Pacritinib) (N=0) | Group VI (Ruxolitinib) (N=0) | Group VII (Idelalisib) (N=0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA | NA
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA | NA
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | NA | NA | NA | NA
Arthritis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA | NA
Hyperleukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA | NA
Blood bilirubin increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA | NA
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA | NA
Short of breath (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA | NA
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA | NA
Troponemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA | NA
Creatinine increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA | NA
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA | NA
Dyspnea (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA | NA
Elevated LFTs (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA | NA
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA | NA
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA | NA
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA | NA
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | NA | NA | NA | NA
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | NA | NA | NA | NA
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | NA | NA | NA | NA
Platelet count decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | NA | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA | NA
White blood cell decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT01620216/Prot_SAP_000.pdf